CLINICAL TRIAL: NCT00879684
Title: A Phase 1, Multicenter, Open-label, Dose-escalation, Safety, Pharmacokinetic, And Pharmacodynamic Trial Of Cvx-060, A Selective Angiopoietin-2 (Ang-2) Binding, Anti-angiogenic Covx-body, In Patients With Advanced Solid Tumors
Brief Title: Safety And PK Study Of CVX-060 In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1131002; CVX-060-101 (Other: Alias Study Number)
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Solid Tumors; Neoplasms; Carcinoma; Cancer; Malignancy
Keywords: Phase 1; Tumors; CVX-060
MeSH Terms: conditions — Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: CVX-060

INTERVENTIONS:
Biological: CVX-060 — Weekly, intravenous dose

SUMMARY:
The purpose of this study is to determine the safety and tolerability of CVX-060 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed advanced solid tumors unresponsive to currently available therapies or for which there is no standard therapy.
* Adequate coagulation, liver, and renal function.
* Candidate for DCE-MRI evaluations.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.

Exclusion Criteria:

* Evidence of significant bleeding problems.
* History of certain gastrointestinal problems including fistula and abscess.
* Chronic, uncontrolled hypertension.
* Patients with any history of primary or metastatic tumor involvement of the brain or with tumors that encase great vessels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Scottsdale Medical Imaging, Ltd., Scottsdale, Arizona
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Premiere Oncology, A Medical Corporation, Santa Monica, California
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1131002&StudyName=Safety%20And%20PK%20Study%20Of%20CVX-060%20In%20Patients%20With%20Advanced%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Groups:
- CVX-060 0.3 mg/kg (Stage 1): CVX-060 0.3 milligram per kilogram (mg/kg) of body weight intravenous infusion administered once-weekly in a 4-week cycle in dose escalation stage (Stage 1).
- CVX-060 1 mg/kg (Stage 1): CVX-060 1 mg/kg of body weight intravenous infusion administered once-weekly in a 4-week cycle in dose escalation stage (Stage 1).
- CVX-060 3 mg/kg (Stage 1): CVX-060 3 mg/kg of body weight intravenous infusion administered once-weekly in a 4-week cycle in dose escalation stage (Stage 1).
- CVX-060 6 mg/kg (Stage 1): CVX-060 6 mg/kg of body weight intravenous infusion administered once-weekly in a 4-week cycle in dose escalation stage (Stage 1).
- CVX-060 12 mg/kg (Stage 1): CVX-060 12 mg/kg of body weight intravenous infusion administered once-weekly in a 4-week cycle in dose escalation stage (Stage 1).
- CVX-060 15 mg/kg (Stage 1): CVX-060 15 mg/kg of body weight intravenous infusion administered once-weekly in a 4-week cycle in dose escalation stage (Stage 1).
- CVX-060 15 mg/kg (Stage 2): CVX-060 15 mg/kg of body weight intravenous infusion administered once-weekly in a 4-week cycle in expanded cohort stage (Stage 2) after completion of dose escalation stage.
Period: Stage 1: Dose Escalation
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 2)
Started | 3 | 3 | 3 | 6 | 3 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 6 | 3 | 3 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 3 | 0 | 4 | 3 | 3 | 0
Not completed — Investigator declined participation | 0 | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Stage 2: Expanded Cohort
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 2)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 13
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 11
Not completed — Investigator declined participation | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants in the study who received any study medication.
Groups:
- CVX-060 (Stage 1 and 2): CVX-060 0.3, 1, 3, 6, 12, 15 mg/kg of body weight intravenous infusion in Stage 1 and CVX-060 15 mg/kg of body weight intravenous infusion in Stage 2, administered once-weekly in a 4-week cycle.
Arm/Group | CVX-060 (Stage 1 and 2)
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to CVX-060 was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline (Day 0) up to 30 days after last dose of study medication
Population: Safety population included all enrolled participants in the study who received any study medication.
Measure: Number; unit: participants
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 2)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 13
participants | 2 | 3 | 1 | 2 | 2 | 1 | 2

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: 0 hour (pre-dose) on Day 0 up to Day 7 of cycle 1 (28 days cycle)
Population: Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of CVX-060 and had PK data.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- CVX-060 15 mg/kg (Stage 1 and 2): CVX-060 15 mg/kg of body weight intravenous infusion in both Stage 1 and Stage 2 administered once-weekly in a 4-week cycle.
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1 and 2)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 16
nanogram per milliliter (ng/mL) | 10550 (1358.4) | 22660 (5230.7) | 68280 (11149) | 140300 (28247) | 249600 (58381) | 318600 (66472)

3. Secondary Outcome: Serum Decay Half-Life (t1/2)
Description: Serum decay half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: 0 hour (pre-dose) on Day 0 up to Day 7 of cycle 1 (28 days cycle)
Population: PK analysis set included all participants who received at least 1 dose of CVX-060 and had PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1 and 2)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 16
hours | 138.1 (36.927) | 92.23 (36.229) | 86.83 (25.002) | 115.2 (32.536) | 124.7 (19.009) | 129.9 (51.813)

4. Secondary Outcome: Area Under the Curve From Time Zero to 168 Hours [AUC (0-168)]
Description: AUC (0-168)= Area under the serum concentration versus time curve from time zero (pre-dose) to 168 hours after dosing (Day 7).
Time Frame: 0 hour (pre-dose) on Day 0 up to Day 7 of cycle 1 (28 days cycle)
Population: PK analysis set included all participants who received at least 1 dose of CVX-060 and had PK data.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1 and 2)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 16
nanogram*hour per milliliter (ng*hr/mL) | 1030000 (155260) | 1644000 (606660) | 5259000 (1127200) | 11990000 (3437600) | 23700000 (2254600) | 26410000 (6658800)

5. Secondary Outcome: Apparent Volume of Distribution (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after intravenous infusion dose (Vss) is influenced by the fraction absorbed.
Time Frame: 0 hour (pre-dose) on Day 0 up to Day 7 of cycle 1 (28 days cycle)
Population: PK analysis set included all participants who received at least 1 dose of CVX-060 and had PK data.
Measure: Geometric Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1 and 2)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 16
milliliter per kilogram (mL/kg) | 32.34 (7.8869) | 54.15 (9.4875) | 50.70 (7.9900) | 51.07 (12.451) | 54.58 (5.1033) | 59.67 (12.711)

6. Secondary Outcome: Apparent Clearance (CL)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). Clearance obtained after intravenous infusion dose (apparent clearance) is influenced by the fraction of the dose absorbed.
Time Frame: 0 hour (pre-dose) on Day 0 up to Day 7 of cycle 1 (28 days cycle)
Population: PK analysis set included all participants who received at least 1 dose of CVX-060 and had PK data.
Measure: Geometric Mean (Standard Deviation); unit: (mL/hr)/kg
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1 and 2)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 16
(mL/hr)/kg | 0.1684 (0.02788) | 0.4399 (0.30607) | 0.4225 (0.12469) | 0.3222 (0.10413) | 0.3078 (0.05000) | 0.3483 (0.16529)

7. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax)
Time Frame: 0 hour (pre-dose) on Day 0 up to Day 7 of cycle 1 (28 days cycle)
Population: PK analysis set included all participants who received at least 1 dose of CVX-060 and had PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1 and 2)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 16
hours | 2.35 [1.58 to 2.37] | 1.50 [1.42 to 2.50] | 2.62 [2.50 to 3.37] | 2.54 [1.50 to 7.37] | 2.42 [2.25 to 2.50] | 2.50 [1.50 to 26.0]

8. Secondary Outcome: Recommended Phase 2 Dose (RP2D): Stage 1
Description: RP2D was determined as the highest dose where none out of 3 (0/3) or less than or equal to 1 out of 6 (<=1/6) participants experienced a dose limiting toxicity (DLT) or was determined based on the safety, pharmacokinetic, and pharmacodynamic findings. DLT was first course AE defined based on National Cancer Institute common toxicity criteria for adverse events version 3 (NCI-CTCAE Version 3) as any hematologic or non-hematologic toxicity greater than or equal to (>=) Grade 3.
Time Frame: Baseline (Day 0) up to 42 days after the last dose of study medication
Population: Safety population included all enrolled participants in the study who received any study medication.
Measure: Number; unit: (mg/kg)/week
Groups:
- CVX-060 (Stage 1): All participants who received 0.3, 1, 3, 6, 12, 15 mg/kg intravenous infusion once-weekly in Stage 1. Participants who discontinued treatment at any time were followed for 6 weeks to assess toxicity, pharmacokinetics (elimination half-life), and immunogenicity.
Arm/Group | CVX-060 (Stage 1)
Number analyzed (Participants) | 21
(mg/kg)/week | 15

9. Secondary Outcome: Number of Participants With Anti-CVX-060 Antibodies
Time Frame: Baseline (Day 0) up to 42 days after last dose
Population: Anti-drug antibodies (ADA) analysis set included all participants who received at least 1 dose of CVX-060 and had PK data.
Measure: Number; unit: participants
Groups:
- CVX-060 (Stage 1 and 2): CVX-060 0.3, 1, 3, 6, 12, 15 mg/kg of body weight intravenous infusion in Stage 1 and CVX-060 15 mg/kg of body weight intravenous infusion in Stage 2 administered once-weekly in a 4-week cycle.
Arm/Group | CVX-060 (Stage 1 and 2)
Number analyzed (Participants) | 34
participants | 20

10. Secondary Outcome: Number of Samples From Participants With Anti-CVX-060 Antibodies
Time Frame: Baseline (Day 0) up to 42 days after last dose
Population: as for outcome 9
Measure: Number; unit: samples
Units Other Than Participants: Samples
Arm/Group | CVX-060 (Stage 1 and 2)
Number analyzed (Participants) | 34
Number analyzed (Samples) | 255
samples | 45

11. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: BOR: best response recorded from treatment start until disease progression/recurrence based on Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR): disappearance of all lesions. Partial Response (PR): >=30% decrease in sum of longest diameters (SLDs) of target lesions taking as reference baseline SLDs, associated to non-progressive disease (non-PD) response for non-target (NT) lesions. PD: >=20% increase in SLDs of target lesions taking as reference smallest SLDs since treatment start, or appearance of >=1 new lesion, or unequivocal progression in NT lesions. Stable disease (SD): neither shrinkage for CR/PR nor increase for PD taking as reference smallest SLDs since treatment start. CR and PR had to be confirmed on a follow up imaging assessment >=4 weeks after initial objective documentation of response. SD criteria should be met at least once after start of treatment in a minimum interval of 8 weeks. Participants with >=3 treatments cycles were reported.
Time Frame: Day 0 (predose), assessed every 8 weeks (2 cycles) until disease progression, unacceptable toxicity, or withdrawal for other reasons (up to Week 133)
Population: Safety population included all enrolled participants in the study who received any study medication.
Measure: Number; unit: participants
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 2)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 13
participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 2 | 2 | 1 | 3 | 1 | 1 | 6
  Progressive Disease | 1 | 1 | 0 | 0 | 2 | 2 | 3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CVX-060 0.3 mg/kg (Stage 1) | CVX-060 1 mg/kg (Stage 1) | CVX-060 3 mg/kg (Stage 1) | CVX-060 6 mg/kg (Stage 1) | CVX-060 12 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 1) | CVX-060 15 mg/kg (Stage 2)
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/3 | 3/6 | 0/3 | 0/3 | 3/13
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6 | 3/3 | 3/3 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVX-060 0.3 mg/kg (Stage 1) (N=3) | CVX-060 1 mg/kg (Stage 1) (N=3) | CVX-060 3 mg/kg (Stage 1) (N=3) | CVX-060 6 mg/kg (Stage 1) (N=6) | CVX-060 12 mg/kg (Stage 1) (N=3) | CVX-060 15 mg/kg (Stage 1) (N=3) | CVX-060 15 mg/kg (Stage 2) (N=13)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVX-060 0.3 mg/kg (Stage 1) (N=3) | CVX-060 1 mg/kg (Stage 1) (N=3) | CVX-060 3 mg/kg (Stage 1) (N=3) | CVX-060 6 mg/kg (Stage 1) (N=6) | CVX-060 12 mg/kg (Stage 1) (N=3) | CVX-060 15 mg/kg (Stage 1) (N=3) | CVX-060 15 mg/kg (Stage 2) (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular retrobulbar haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 4
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 0 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 2
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 0 | 2 | 1 | 0 | 2
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 2 | 2 | 1 | 0 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Smear cervix abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suture removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Designation of outcomes as primary, secondary was based on study team's input as study did not specify them as primary or secondary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.